CLINICAL TRIAL: NCT05835869
Title: Electrophysiological and Morphofunctional Changes of Retina and Choroid Vascularization After Carotid Endarterectomy, a Pilot Study
Brief Title: Chorioretinal Vascularization and Electrophysiological Changes After Carotid Revascularization
Acronym: CAS-AOCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5532
Record Dates: First submitted 2023-04-19; First posted 2023-04-28 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-04

CONDITIONS: Carotid Stenosis
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study population (Experimental)
  Interventions: Diagnostic Test: Optical coherence tomography angiography and pattern electroretinogram

INTERVENTIONS:
Diagnostic Test: Optical coherence tomography angiography and pattern electroretinogram — Optical coherence tomography angiography is an infrared eye scan that analyzes retinal vascularization and anatomy

SUMMARY:
The aim of the study is to evaluate changes in retinal function by means of electro-functional examinations of the retina and to associate them with any changes in chorioretinal vascular density occurring in the ipsilateral eye after carotid revascularization surgery.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years old
* Carotid stenosis diagnosis with indication to perform carotid endarterectomy
* informed consent form signing

Exclusion Criteria:

* age <18 years old
* recurrent intraocular inflammation
* retinal disease
* optic neuropathy, optic nerve drusen, opacity of the dioptric means in the pre- or post-operative period that prevents the acquisition of high-resolution images
* unstable fixation
* spheric refractive error > +/- 6 D spheric and/or +/- 3 D cylinder
* history of prior ocular surgery
* refusal of signing informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Functional retinal changes | 1 week and 3 months
  To evaluate rate of pattern electroretinography/pattern visual evoked potential improvement in both eyes before and after carotid endarterectomy

SECONDARY OUTCOMES:
Retinal vascular density changes | 1 week and 3 months
  To evaluate rate of chorioretinal vascular density improvement trough angiographic optical coherence tomography before and after carotid endarterectomy

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Baldascino, MD, Principal Investigator — Policlinico Agostino Gemelli IRRCS
Locations (1):
- Policlinico Agostino Gemelli IRCCS, Roma, RM, Italy